CLINICAL TRIAL: NCT00963326
Title: Morphological and Molecular Characterization of Tumors of the Aero-digestive Tract in Patients Who Have no Risk Factors Such as Alcohol, Smoking, or Occupation
Brief Title: Study of Blood and Tissue Samples From Patients With Larynx Cancer, Pharynx Cancer, or Oral Cavity Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000635996; COL-CARIO; 2007-11; INCA-RECF0897; ID-RCB-2008-A00300-55
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent verrucous carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent verrucous carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood and tissue samples from patients with larynx cancer, pharynx cancer, or oral cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Characterize, morphologically and molecularly, squamous cell carcinoma of the larynx, pharynx, or oral cavity in patients without high-risk factors, such as alcohol consumption, smoking, or occupation.

Secondary

* Study the impact parameters of morphology, molecular characteristics, and genomics on disease-free survival and overall survival of these patients.
* Study the impact parameters of morphological, molecular, and genomic control in the tumor.
* Assess, in advanced tumors, the risk of heterogeneity of morphological, molecular, and genomic control in the tumor.

OUTLINE: This is a multicenter study.

Blood, tumor tissue, and healthy tissue samples are collected before treatment begins.

Patients are followed up every 3 months for 2 years (additional biopsies may be collected).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the larynx, pharynx, or oral cavity
* No risk factors of alcohol consumption, smoking, or occupational hazards such as asbestos, hydrocarbons, paints, nickel, stone dust, or wood dust.

  * Must be a life-time non-smoker, not a former smoker
* Measurable disease by RECIST criteria

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* No other serious concomitant medical conditions precluding general anesthesia
* No psychological, familial, social, or geographical reasons that would preclude follow up

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Lefebvre, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France